CLINICAL TRIAL: NCT05101785
Title: Articaine 4% Efficacy and Safety in Extraction and Pulpotomy of Primary Molars of Children Below the Age of Four Years.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Mahmoud Ahmed Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Mahmoud Ahmed Mahmoud, Lecturer, Minia University
Organization: Minia University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 3081
Record Dates: First submitted 2021-10-28; First posted 2021-11-01 (Actual); Last update posted 2021-11-01 (Actual); Status verified 2021-10

CONDITIONS: Pain; Behavior
MeSH Terms: conditions — Pain; Behavior | interventions — Epinephrine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lidocaine (Active Comparator): Lidocain hydrochloride 2 %with epinephrine 1:100000
  Interventions: Drug: Lidocain hydrochloride 2 % with epinephrine
- Articaine (Experimental): Articaine chloride 4% with epinephrine 1:100000
  Interventions: Drug: Articaine chloride 4% with epinephrine

INTERVENTIONS:
Drug: Lidocain hydrochloride 2 % with epinephrine — Local anesthesia infilteration in children
  Arms: Lidocaine
Drug: Articaine chloride 4% with epinephrine — Articaine chloride 4% with epinephrine
  Arms: Articaine

SUMMARY:
compare the anaesthetic efficacy and safety for pain and behaviour for extraction or pulp therapy in primary molars in young children below four years old using 4% articaine and 2% lidocaine local anesthetics.

ELIGIBILITY:
Inclusion Criteria:

* Healthy children
* 3-6 years
* primary molar indicated for pulpotomy
* body weight not less than 15 Kg

Exclusion Criteria:

* Intellectual problem
* sever emotional problems
* previous dental experience
* Medically or mentally compromised children

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 292 (Estimated)
Dates: Start 2021-11-01 (Estimated); Primary Completion 2022-09-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
Intra and post operative pain | 30-60 minutes
  Evaluate pain during injection and treatment using FLACC (face,legs,activity, cry, consolabolity) scale
Behavior | 30-60 minutes
  Evaluate child behavior using frankl scale during treatment
Blood pressure | 30-60 minutes
  Vital signs
Heart rate | 30-60 minutes
  Vital signs
Respiratory rate measuring during treatment | 30-60 minutes
  Vital signs